CLINICAL TRIAL: NCT06427031
Title: A Multi-center, Randomized, Double-blinded, Active Control, Parallel, Phase 3 Trial to Evaluate the Efficacy and Safety of TJO-083 in Dry Eye Diseases Patients
Brief Title: Comparing Efficacy and Safety of TJO-083 in Dry Eye Diseases Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJO-083-A03
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Double-blind, Active control for Evaluating the Efficacy and Safety of the test drug(TJO-083) Compared with the control drug in Dry Eye Sydrome
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TJO-083 (Experimental): TJO-083 : 1 drop 3 times a day
  Interventions: Drug: TJO-083
- Diquas-s Ophthalmic solution 3% 0.4mL (Active Comparator): 1 drop 6 times a day
  Interventions: Drug: Diquafosol ophthalmic sodium solution 3%

INTERVENTIONS:
Drug: TJO-083 — Diquafosol ophthalmic sodium solution, 1 drop 3 times a day
  Arms: TJO-083
Drug: Diquafosol ophthalmic sodium solution 3% — Diquafosol ophthalmic sodium solution, 1 drop 6 times a day
  Arms: Diquas-s Ophthalmic solution 3% 0.4mL

SUMMARY:
In patients with dry eye syndrome, the test drug(TJO-083) or the control drug is administered for 12 weeks, and the corneal staining of each group would be evaluated. The purpose of this clinical Study is to demonstrate that the test drug is not clinically inferior to the control drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 or over
* Has dry eye symptoms (minimum 3 months)
* Screening both eyes, the corrected visual acuity is 0.2 or more
* Written informed consent to participate in the trial

Exclusion Criteria:

* The patients who treated with topical NSAIDs/hyaluronate sodium ophthalmic solutions within 2 weeks of randomized visits.
* The patients with systemic or ocular disorders affecting the test results(ocular surgery, trauma, or disease) within 2 months of screening visits.
* Intraocular pressure(IOP)> 21 mmHg
* Patients with contact lens

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Corneal Staining at Week 4 | Baseline and Week 4
  Change from Baseline in corneal staining using blue fluorescein staining procedure at Week 4.

SECONDARY OUTCOMES:
Change From Baseline in Corneal Staining at Week 8, 12 | Baseline and Week 8 and 12
  Change from Baseline in corneal staining using blue fluorescein staining procedure at Week 8, 12.
Change From Baseline in Conjunctival Staining at Week 4, 8 and 12 | Baseline and Week 4, 8 and 12
  Change From Baseline in Conjunctival Staining using Rose Bengal staining procedure at Week 4, 8 and 12
Change From Baseline in Non-anesthetic Schirmer Test at Week 4, 8, 12 | Baseline and Week 4, 8 and 12
  The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac.

CONTACTS AND LOCATIONS:
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No